CLINICAL TRIAL: NCT06249880
Title: Pediatric Normative Markerless Movement Analysis Data Collection Project
Brief Title: Pediatric Normative Markerless Movement Analysis
Status: Recruiting | Type: Observational
Sponsor: MultiCare Health System Research Institute (Other)
Responsible Party: Sponsor
Other Study IDs: #2023/11/2
Record Dates: First submitted 2024-01-24; First posted 2024-02-08 (Actual); Last update posted 2024-02-16 (Actual); Status verified 2024-02

CONDITIONS: Pediatric ALL; Adolescent
Keywords: Motion Analysis; Kinetics; Kinematics
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — Observation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Normative: 40 neurotypical pediatric subjects
  Interventions: Other: Observation

INTERVENTIONS:
Other: Observation — This project seeks to recruit 20 male and 20 female typically developing individuals, between the ages of 3 and 25 years of age. Non-invasive measurements of movement patterns (motion analysis and force plate data) will be collected during bipedal gait.

SUMMARY:
The objective of this project is to collect baseline data from a normative population of children that gender and age matches the population of patients expected to be treated by Mary Bridge Children's Research & Movement Lab. This project seeks to recruit 20 male and 20 female typically developing individuals, between the ages of 3 and 25 years of age. Non-invasive measurements of movement patterns (motion analysis and force plate data) will be collected during bipedal gait.

ELIGIBILITY:
Inclusion Criteria:

* Age: 3-25 years of age (with 3 and 25 year olds considered for inclusion).
* Ambulate independently and without the use of assistive devices or orthoses.
* Willing and interested in participating.

Exclusion Criteria:

* Neuromuscular disorders such as cerebral palsy, muscular dystrophy, myotonic dystrophy, spinal muscular atrophy, peripheral neuropathy, or other generalized muscle and/or nerve issues.
* Evidence of developmental delays, muscle weakness, decreased muscle tone, joint stiffness, muscle or bone deformity.
* Currently using or has a history of using assistive technology devices, bracing/orthoses, manual or powered mobility equipment.
* History of premature birth.
* Currently or has a history of taking medication or pharmaceutical treatment related to musculoskeletal side-effects/scenario/diagnosis.

Ages: 3 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Subjects will be recruited from the regional community, including convenience sample of children. Subjects will be recruited by word of mouth, posted flyers, and advertised through the RML website and MB social media.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2024-02-14 (Estimated); Primary Completion 2025-02-14 (Estimated); Study Completion 2025-02-14 (Estimated)

PRIMARY OUTCOMES:
Observation-based movement analyses | Baseline
  The purpose of this normative data collection study is to collect baseline data from a normative population of children/adolescents using force plates and 3D markerless motion capture. Together these are used to calculate a normative range of body position and joint angles (kinematics), as well as joint loads and ground reaction forces (kinetics) during prescribed activities.

CONTACTS AND LOCATIONS:
Locations (1):
- Mary Bridge Children's Therapy Unit - Research & Movement Lab, Puyallup, Washington, United States